CLINICAL TRIAL: NCT05409716
Title: Comparison Between Compressive Elastic Dressing and Hemostatic TR Band Following Cardiac Intervention Utilizing the Radial Technique: A Randomized Controlled Trial
Brief Title: Compressive Elastic Dressing Versus TR Band
Acronym: Band Vs Gauze
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: An-Najah National University (Other)
Responsible Party: Principal Investigator, Yunis Daralammouri, Assistant Professor, An-Najah National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TR-Band Vs Gauze Swab
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Angina, Unstable; Angina, Stable; Acute Coronary Syndrome; STEMI; NSTEMI; Ischemic Heart Disease; Atherosclerotic Cardiovascular Disease; Chest Pain; Non ST Elevation Myocardial Infarction
Keywords: Radial approach; Wristband; TR Band; compressive dressing; cardiac catheterization; radial artery; safeguard; randomized controlled trial
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Angina, Unstable; Angina, Stable; Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Myocardial Ischemia; Atherosclerosis; Chest Pain | interventions — Hemostasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients enrolled to the study were randomized into TR Band or compressive dressing groups. Care providers operated on patients and investigators collected their data during and after the operation. The independent variable - Hemostasis technique (TR Band or compressive dressing ) - was coded into X or Z groups, then data was sent to the outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressive Elastic dressing (Experimental): Patients who received compressive elastic dressing as a hemostasis technique after coronary angiography using radial approach.
  Interventions: Procedure: Compressive Elastic dressing for hemostasis in cardiac procedure using radial approach
- wristband TR Band (Active Comparator): Patients who received wristband TR Band as a hemostasis technique after coronary angiography using radial approach.
  Interventions: Procedure: Wristband TR band for hemostasis in cardiac procedure using radial approach

INTERVENTIONS:
Procedure: Compressive Elastic dressing for hemostasis in cardiac procedure using radial approach — Following cardiac procedure using radial approach, compressive elastic dressing, standardized as 13 threads gauze overlapped, opened, longitudinally pleated once and wrapped, making a 5-cm long cylinder, 1-cm in height, fixed with elastic crepe bandage was used to achieve hemostasis.
  Arms: Compressive Elastic dressing
Procedure: Wristband TR band for hemostasis in cardiac procedure using radial approach — Following cardiac procedure using radial approach, hemostatic wristband TR BandR (Terumo Corporation, Tokyo, Japan) was utilized was used to achieve hemostasis.
  Arms: wristband TR Band

SUMMARY:
Radial approach is widely established in cardiac diagnostic and therapeutic treatments. It has been shown to decrease bleeding, vascular problems, and mortality rates when compared to the femoral approach. It also offers better comfort to patients through early mobility and lowers hospital expenses.

Previously, there were no specific devices for radial artery hemostasis. Many different types of dressings were used in various hospitals with no standardization. This raises the question of whether specific devices surpass dressings in terms of patient comfort, time required to maintain hemostasis, and vascular complications.

The primary goal of this study was to examine the effectiveness of compression dressings and hemostatic wristbands on patients undergoing cardiac procedures via radial approach in terms of patient comfort, time required to maintain hemostasis, and vascular problems.

The hemostatic wristband TR BandR (Terumo Corporation, Tokyo, Japan) was utilized in one group, while compressive elastic dressing, standardized as 13 threads gauze overlapped, opened, longitudinally pleated once and wrapped, making a 5-cm long cylinder, 1-cm in height, was used in the other.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients who agree to participate in the study and sign the consent form.
* Patients with an indication for coronary catheterization
* Clinically stable patients
* Patients with palpable pulses on at least one of the radial arteries.

Exclusion Criteria:

* Patients who are hemodynamically unstable (systolic blood pressure less 90mmhg)
* Patients with radial AV shunt for hemodialysis
* Patients with previous CABG using radial artery
* Patients with Renaud phenomenon or lymphedema
* Patients who had vascular problems at the puncture site before the hemostasis process started.
* Failure to obtain radial access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Compression "hemostasis" time | Up to 240 minutes after placement
  The time from the placement of the hemostatic Wristband or Compressive dressing until its removal (when there's no blood oozing after removal), measured by minutes.
Number of patient with Hematoma and Grade of hematoma | Within 24 hours after the procedure
  It is defined by EASY hematoma scale.

SECONDARY OUTCOMES:
Number of patient with Radial artery occlusion | Within 24 hours after the procedure
  Radial artery patency was checked by evaluating radial pulse, capillary refill, hand color, temperature, and assessing the puncture site and hand for any hematoma or bleeding. In the event of an access site hematoma or any other ischemia sign, the patient will be sent to the radiology department for further assessment with radial artery Doppler.
Ischemic changes to the hand | Within 24 hours after the procedure
  It is noted by clinical features of pallor, absence of pulse, pain, cold, paresthesia or paralysis.
Post-procedural pain | Within 24 hours after the procedure
  Assessed by numerical rating scale (NRS) for pain, which is an 11 point subjective scale (0-10) where 0 refers for no pain, 1-3 for mild pain, 4-6 for moderate pain and 7-10 for severe pain.
Number of patient with Radial Artery Occlusion on follow up | After 4 weeks of the procedure.
  Radial artery patency was checked by evaluating radial pulse and Doppler Ultrasonography.
Patient satisfaction of the used compression methode Assessed by Likert scale for satisfaction | Within 24 hrs
  Assessed by Likert scale for satisfaction , which is a 5 point subjective scale (1-5) where 1 refers for Not at all satisfied , 2 for slightly satisfied , 3 for moderately satisfied, 4 for Very satisfied and 5 for Extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Yunis A Daralammouri, Principal Investigator — An-Najah National University
Locations (2):
- Palestinian Territories (2):
  - An-Najah National University Hospital, Nablus, West Bank
  - An-Najah National University Hospital, Nablus